CLINICAL TRIAL: NCT01513239
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy, Safety and Tolerability of a Single Infusion of MK-6072 (Human Monoclonal Antibody to Clostridium Difficile Toxin B), and MK-3415A (Human Monoclonal Antibodies to Clostridium Difficile Toxin A and B) in Patients Receiving Antibiotic Therapy for Clostridium Difficile Infection (MODIFY II)
Brief Title: A Study of MK-6072 and MK-3415A in Participants Receiving Antibiotic Therapy for Clostridium Difficile Infection (MK-3415A-002)
Acronym: MODIFY II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3415A-002; 132231 (Registry Identifier: JAPIC-CTI); 2011-004994-94 (EudraCT Number)
Record Dates: First submitted 2012-01-16; First posted 2012-01-20 (Estimated); Results first posted 2016-12-15 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Clostridium Difficile Infection
Keywords: Clostridium difficile; Clostridium difficile infection (CDI); recurrent Clostridium difficile; vancomycin; metronidazole; monoclonal antibody
MeSH Terms: conditions — Clostridium Infections | interventions — bezlotoxumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- MK-6072 + SOC (Experimental): Single intravenous (IV) infusion of 10 mg/kg MK-6072 + Standard of Care (SOC) for CDI
  Interventions: Biological: MK-6072; Drug: SOC
- MK-3415A + SOC (Experimental): Single IV infusion of 10 mg/kg MK-3415A + SOC for CDI
  Interventions: Biological: MK-3415A; Drug: SOC
- Placebo + SOC (Placebo Comparator): Normal saline IV infusion (0.9% sodium chloride) + SOC for CDI
  Interventions: Biological: Placebo; Drug: SOC

INTERVENTIONS:
Biological: MK-6072 — Single IV infusion of MK-6072 (10 mg/kg of monoclonal antibody to C. difficile Toxin B)
  Arms: MK-6072 + SOC
Biological: MK-3415A — Single IV infusion of MK-3415A (10 mg/kg of monoclonal antibody to C. difficile Toxin A and 10 mg/kg of monoclonal antibody to C. difficile Toxin B)
  Arms: MK-3415A + SOC
Biological: Placebo — Single IV infusion of normal saline (0.9% sodium chloride)
  Arms: Placebo + SOC
Drug: SOC — SOC for CDI will be prescribed for 10 to 14 days and can begin on the day of study drug infusion; but the first dose must have been administered prior to or within a few hours following study drug infusion. SOC is defined as the receipt of oral metronidazole, oral vancomycin, IV metronidazole concurrent with oral vancomycin, oral fidaxomicin, or oral fidaxomicin concurrent with IV metronidazole.

SUMMARY:
MK-3415A is the combination of monoclonal antibodies to Clostridium (C.) difficile toxin A (MK-3415) and toxin B (MK-6072). This study will investigate whether: 1) treatment with MK-6072 or MK-3415A in addition to standard of care (SOC) antibiotic therapy will decrease Clostridium Difficile Infection (CDI) recurrence compared with placebo; and 2) MK-6072 and MK-3415A will be generally well tolerated in participants receiving SOC therapy for CDI compared with placebo.

DETAILED DESCRIPTION:
An extended 9-month follow-up to assess for CDI recurrence through Month 12 will be conducted in a subset of participants.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a diagnosis of CDI defined as: a) presence of diarrhea (passage of 3 or more loose stools in 24 or fewer hours); and b) positive test for toxigenic C. difficile from a stool collected no more than 7 days before study infusion.
* Participant is receiving SOC therapy (i.e., oral metronidazole, oral vancomycin, IV metronidazole concurrent with oral vancomycin, oral fidaxomicin, or oral fidaxomicin concurrent with IV metronidazole) for CDI.
* Participant is highly unlikely to become pregnant or to impregnate a partner by meeting at least one of the following criteria: a) females not of reproductive potential (i.e., one who has either (1) reached natural menopause, defined as 6 months of spontaneous amenorrhea with serum follicle stimulating hormone [FSH] levels in the postmenopausal range, or 12 months of spontaneous amenorrhea not including cases with an underlying disease, such as anorexia nervosa, that causes amenorrhea; (2) 6 weeks post surgical bilateral oophorectomy with or without hysterectomy; or (3) bilateral tubal ligation); or b) participants of reproductive potential who agree to remain abstinent or use (or have their partner use) two acceptable methods of birth control (i.e., intrauterine device [IUD], diaphragm with spermicide; contraceptive sponge, condom, vasectomy and any registered and marketed hormonal contraceptives that contain an estrogen and/or progestational agent including oral, subcutaneous, intrauterine, or intramuscular agents) starting at enrollment and throughout the 12-week study.

Exclusion Criteria:

* Participant with an uncontrolled chronic diarrheal illness such that their normal 24-hour bowel movement habit is 3 or more loose stools.
* Participant with planned surgery for CDI within 24 hours.
* Female participant with a positive pregnancy test in the 48 hours before infusion and pre-menopausal females who are not sterilized and therefore have the potential to bear a child who are unwilling to undergo pregnancy testing.
* Female participant breast feeding or planning to breast feed before completion of the 12-week study.
* Female participant planning to donate ova before completion of the 12-week study and male participants planning to impregnate or donate sperm before completion of the 12-week study.
* Participant has previously participated in this study, has previously received MK-3415 or MK-6072 (either alone or in combination), has received a C. difficile vaccine, or has received another experimental monoclonal antibody against C. difficile toxin A or B.
* Participant plans to donate blood and/or blood products within 6 months after infusion.
* Participant has received immune globulin within 6 months before infusion or is planning to receive immune globulin before completion of the 12-week study.
* Treatment with SOC therapy is planned for longer than 14 days.
* Participant has received more than a 24-hour regimen of cholestyramine, colestimide, rifaximin, or nitazoxanide within 14 days before infusion or plans to receive these medication before completion of the 12-week study period.
* Participant plans to take medications that are given to decrease gastrointestinal peristalsis, such as loperamide (Imodium™) or diphenoxylate hydrochloride/atropine sulfate (Lomotil™) any time during the 14 days after infusion. Participants receiving opioid medications at the onset of diarrhea may be included if they are on a stable dose or if there is anticipation of a dose decrease or cessation of use.
* Participant plans to take the probiotic Saccaromyces boulardii or plans to receive fecal transplantation therapy, or any other therapies that have been demonstrated to decrease CDI recurrence at any time after infusion (Day 1) and through completion of the 12-week study period.
* Participant has received another investigational study agent within the past 30 days or is currently participating in or scheduled to participate in any other clinical study with an investigational agent during the 12-week study.
* Participant is not expected to survive for 72 hours.
* Participant has any other condition that, in the opinion of the investigator, would jeopardize the safety or rights of the participant, would make it unlikely for the participant to complete the study, or would confound the results of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1203 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2015-05-22 (Actual); Study Completion 2015-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] de Almeida C, Wong M, Kleijn HJ, Wrishko RE. Predicted Bezlotoxumab Exposure in Patients Who Have Received a Hematopoietic Stem Cell Transplant. Clin Ther. 2023 Apr;45(4):356-362. doi: 10.1016/j.clinthera.2023.02.006. Epub 2023 Mar 9. PMID 36906440
- [Derived] Zhang H, Mehrotra DV, Shen J. AWOT and CWOT for genotype and genotype-by-treatment interaction joint analysis in pharmacogenetics GWAS. Bioinformatics. 2023 Jan 1;39(1):btac834. doi: 10.1093/bioinformatics/btac834. PMID 36661328
- [Derived] Bouza E, Cornely OA, Ramos-Martinez A, Plesniak R, Ellison MC, Hanson ME, Dorr MB. Analysis of C. difficile infection-related outcomes in European participants in the bezlotoxumab MODIFY I and II trials. Eur J Clin Microbiol Infect Dis. 2020 Oct;39(10):1933-1939. doi: 10.1007/s10096-020-03935-3. Epub 2020 Jun 6. PMID 32504314
- [Derived] Shen J, Mehrotra DV, Dorr MB, Zeng Z, Li J, Xu X, Nickle D, Holzinger ER, Chhibber A, Wilcox MH, Blanchard RL, Shaw PM. Genetic Association Reveals Protection against Recurrence of Clostridium difficile Infection with Bezlotoxumab Treatment. mSphere. 2020 May 6;5(3):e00232-20. doi: 10.1128/mSphere.00232-20. PMID 32376702
- [Derived] Zhang H, Zhao N, Mehrotra DV, Shen J. Composite Kernel Association Test (CKAT) for SNP-set joint assessment of genotype and genotype-by-treatment interaction in Pharmacogenetics studies. Bioinformatics. 2020 May 1;36(10):3162-3168. doi: 10.1093/bioinformatics/btaa125. PMID 32101275
- [Derived] Cornely OA, Mullane KM, Birch T, Hazan-Steinberg S, Nathan R, Bouza E, Calfee DP, Ellison MC, Wong MT, Dorr MB. Exploratory Evaluation of Bezlotoxumab on Outcomes Associated With Clostridioides difficile Infection in MODIFY I/II Participants With Cancer. Open Forum Infect Dis. 2020 Jan 31;7(2):ofaa038. doi: 10.1093/ofid/ofaa038. eCollection 2020 Feb. PMID 32099847
- [Derived] Goldstein EJC, Citron DM, Gerding DN, Wilcox MH, Gabryelski L, Pedley A, Zeng Z, Dorr MB. Bezlotoxumab for the Prevention of Recurrent Clostridioides difficile Infection: 12-Month Observational Data From the Randomized Phase III Trial, MODIFY II. Clin Infect Dis. 2020 Aug 14;71(4):1102-1105. doi: 10.1093/cid/ciz1151. PMID 31883370
- [Derived] Zeng Z, Zhao H, Dorr MB, Shen J, Wilcox MH, Poxton IR, Guris D, Li J, Shaw PM. Bezlotoxumab for prevention of Clostridium difficile infection recurrence: Distinguishing relapse from reinfection with whole genome sequencing. Anaerobe. 2020 Feb;61:102137. doi: 10.1016/j.anaerobe.2019.102137. Epub 2019 Dec 14. PMID 31846705
- [Derived] Kelly CP, Poxton IR, Shen J, Wilcox MH, Gerding DN, Zhao X, Laterza OF, Railkar R, Guris D, Dorr MB. Effect of Endogenous Clostridioides difficile Toxin Antibodies on Recurrence of C. difficile Infection. Clin Infect Dis. 2020 Jun 24;71(1):81-86. doi: 10.1093/cid/ciz809. PMID 31628838
- [Derived] Montgomery DL, Matthews RP, Yee KL, Tobias LM, Dorr MB, Wrishko RE. Assessment of Bezlotoxumab Immunogenicity. Clin Pharmacol Drug Dev. 2020 Apr;9(3):330-340. doi: 10.1002/cpdd.729. Epub 2019 Aug 14. PMID 31411386
- [Derived] Basu A, Prabhu VS, Dorr MB, Golan Y, Dubberke ER, Cornely OA, Heimann SM, Pedley A, Xu R, Hanson ME, Marcella S. Bezlotoxumab Is Associated With a Reduction in Cumulative Inpatient-Days: Analysis of the Hospitalization Data From the MODIFY I and II Clinical Trials. Open Forum Infect Dis. 2018 Nov 15;5(11):ofy218. doi: 10.1093/ofid/ofy218. eCollection 2018 Nov. PMID 30460321
- [Derived] Yee KL, Kleijn HJ, Kerbusch T, Matthews RP, Dorr MB, Garey KW, Wrishko RE. Population Pharmacokinetics and Pharmacodynamics of Bezlotoxumab in Adults with Primary and Recurrent Clostridium difficile Infection. Antimicrob Agents Chemother. 2019 Jan 29;63(2):e01971-18. doi: 10.1128/AAC.01971-18. Print 2019 Feb. PMID 30455246
- [Derived] Kelly CP, Wilcox MH, Glerup H, Aboo N, Ellison MC, Eves K, Dorr MB. Bezlotoxumab for Clostridium difficile Infection Complicating Inflammatory Bowel Disease. Gastroenterology. 2018 Oct;155(4):1270-1271. doi: 10.1053/j.gastro.2018.06.080. Epub 2018 Sep 15. No abstract available. PMID 30227108
- [Derived] Prabhu VS, Cornely OA, Golan Y, Dubberke ER, Heimann SM, Hanson ME, Liao J, Pedley A, Dorr MB, Marcella S. Thirty-Day Readmissions in Hospitalized Patients Who Received Bezlotoxumab With Antibacterial Drug Treatment for Clostridium difficile Infection. Clin Infect Dis. 2017 Oct 1;65(7):1218-1221. doi: 10.1093/cid/cix523. PMID 30060024
- [Derived] Birch T, Golan Y, Rizzardini G, Jensen E, Gabryelski L, Guris D, Dorr MB. Efficacy of bezlotoxumab based on timing of administration relative to start of antibacterial therapy for Clostridium difficile infection. J Antimicrob Chemother. 2018 Sep 1;73(9):2524-2528. doi: 10.1093/jac/dky182. PMID 29788418
- [Derived] Gerding DN, Kelly CP, Rahav G, Lee C, Dubberke ER, Kumar PN, Yacyshyn B, Kao D, Eves K, Ellison MC, Hanson ME, Guris D, Dorr MB. Bezlotoxumab for Prevention of Recurrent Clostridium difficile Infection in Patients at Increased Risk for Recurrence. Clin Infect Dis. 2018 Aug 16;67(5):649-656. doi: 10.1093/cid/ciy171. PMID 29538686
- [Derived] Wilcox MH, Gerding DN, Poxton IR, Kelly C, Nathan R, Birch T, Cornely OA, Rahav G, Bouza E, Lee C, Jenkin G, Jensen W, Kim YS, Yoshida J, Gabryelski L, Pedley A, Eves K, Tipping R, Guris D, Kartsonis N, Dorr MB; MODIFY I and MODIFY II Investigators. Bezlotoxumab for Prevention of Recurrent Clostridium difficile Infection. N Engl J Med. 2017 Jan 26;376(4):305-317. doi: 10.1056/NEJMoa1602615. PMID 28121498

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male and female participants 18 years of age or older, diagnosed with Clostridium difficile infection (CDI) and receiving Standard of Care (SOC) therapy were recruited for this trial.
Groups:
- MK-3415A + SOC: Single intravenous (IV) infusion of 10 mg/kg MK-3415A + SOC for CDI
- MK-6072 + SOC: Single IV infusion of 10 mg/kg MK-6072 + SOC for CDI
- MK-3415A + SOC 9-ME: 9 Month Extension (9-ME) for participants treated with a single IV infusion of 10 mg/kg MK-3415A + SOC
- MK-6072 + SOC 9-ME: 9-ME for participants treated with a single IV infusion of 10 mg/kg MK-6072 + SOC
- Placebo + SOC 9-ME: 9-ME for participants treated with Placebo
Period: Period 1: Main Phase
Arm/Group | MK-3415A + SOC | MK-6072 + SOC | Placebo + SOC | MK-3415A + SOC 9-ME | MK-6072 + SOC 9-ME | Placebo + SOC 9-ME
Started | 397 (Randomized participants) | 407 (Randomized participants) | 399 (Randomized participants) | 0 | 0 | 0
Treated | 391 (Treated participants) | 396 (Treated participants) | 381 (Treated participants) | 0 | 0 | 0
All Participants as Treated | 390 (One participant randomized to receive MK-3415A (MK-3415 plus MK-6072) received only MK-3415) | 396 (Treatment actually received) | 381 (Treatment actually received) | 0 | 0 | 0
Completed | 322 | 337 | 311 | 0 | 0 | 0
Not Completed | 75 | 70 | 88 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 2 | 0 | 0 | 0
Not completed — Death | 29 | 22 | 32 | 0 | 0 | 0
Not completed — Lost to Follow-up | 11 | 10 | 6 | 0 | 0 | 0
Not completed — Physician Decision | 4 | 4 | 4 | 0 | 0 | 0
Not completed — Protocol Violation | 2 | 2 | 2 | 0 | 0 | 0
Not completed — Technical Problems | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 27 | 29 | 42 | 0 | 0 | 0
Period: Period 2: 9 Month Extension Phase
Arm/Group | MK-3415A + SOC | MK-6072 + SOC | Placebo + SOC | MK-3415A + SOC 9-ME | MK-6072 + SOC 9-ME | Placebo + SOC 9-ME
Started | 0 | 0 | 0 | 112 | 100 | 83
Completed | 0 | 0 | 0 | 102 | 90 | 78
Not Completed | 0 | 0 | 0 | 10 | 10 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 5 | 3 | 2
Not completed — Death | 0 | 0 | 0 | 2 | 5 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Technical Problems | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All Randomized Participants
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-3415A + SOC | MK-6072 + SOC | Placebo + SOC | Total
Number analyzed (Participants) | 397 | 407 | 399 | 1203
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.9 (17.3) | 62.6 (17.5) | 64.3 (16.4) | 64.2 (17.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 216 | 220 | 239 | 675
  Male | 181 | 187 | 160 | 528

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With CDI Recurrence
Description: CDI recurrence is defined as the development of a new episode of diarrhea (3 or more loose stools in 24 or fewer hours) and a positive lab stool test (local or central) for toxigenic C. difficile after clinical cure of the initial CDI episode. Clinical cure is defined as no diarrhea [2 or fewer loose stools per 24 hours] for 2 consecutive days following completion of SOC therapy for the initial CDI episode in participants who received =< 14 day regimen.
Time Frame: 12 weeks
Population: The (Full Analysis Set) FAS population consisting of all randomized participants with participants excluded for the failure to receive infusion of study medication; for lack of a positive local stool test for toxigenic C. difficile; or for failure to receive protocol defined standard of care therapy within a 1 day window of the infusion.
Measure: Number; unit: Percentage of participants
Arm/Group | MK-3415A + SOC | MK-6072 + SOC | Placebo + SOC
Number analyzed (Participants) | 390 | 395 | 378
Percentage of participants | 14.9 | 15.7 | 25.7
Statistical Analysis 1: Comparison: MK-3415A + SOC vs Placebo + SOC; Test type: Superiority or Other; p < 0.0001, Miettinen and Nurminen — One sided p-value based on the Miettinen and Nurminen method stratified by SOC therapy (metronidazole vs. vancomycin vs. fidaxomicin) and hospitalization status (inpatient vs. outpatient); Adjusted Difference = -10.7, 95% CI 2-sided [-16.4 to -5.1] — MK-3415A + SOC minus Placebo + SOC
Statistical Analysis 2: Comparison: MK-6072 + SOC vs Placebo + SOC; Test type: Superiority or Other; p = 0.0003, Miettinen and Nurminen — [p-value comment as in outcome 1, analysis 1]; Adjusted Difference = -9.9, 95% CI 2-sided [-15.5 to -4.3] — MK-6072 + SOC minus Placebo + SOC
Statistical Analysis 3: Comparison: MK-3415A + SOC vs MK-6072 + SOC; Test type: Superiority or Other; p = 0.3718, Miettinen and Nurminen — [p-value comment as in outcome 1, analysis 1]; Adjusted Difference = -0.8, 95% CI 2-sided [-5.9 to 4.2] — MK-3415A + SOC minus MK-6072 + SOC

2. Secondary Outcome: Percentage of Participants With Global Cure
Description: Global cure is defined as the clinical cure of the initial CDI episode with no CDI recurrence through Week 12. Clinical cure is defined as no diarrhea [2 or fewer loose stools per 24 hours] for 2 consecutive days following completion of SOC therapy for the initial CDI episode in participants who received =< 14 day regimen.
Time Frame: 12 weeks
Population: The FAS population consisting of all randomized participants with participants excluded for the failure to receive infusion of study medication; for lack of a positive local stool test for toxigenic C. difficile; or for failure to receive protocol defined standard of care therapy within a 1 day window of the infusion.
Measure: Number; unit: Percentage of participants
Arm/Group | MK-3415A + SOC | MK-6072 + SOC | Placebo + SOC
Number analyzed (Participants) | 390 | 395 | 378
Percentage of participants | 57.4 | 66.8 | 52.1
Statistical Analysis 1: Comparison: MK-3415A + SOC vs Placebo + SOC; Test type: Superiority or Other; p = 0.0722, Miettinen and Nurminen — [p-value comment as in outcome 1, analysis 1]; Adjusted Difference = 5.2, 95% CI 2-sided [-1.8 to 12.2] — MK-3415A + SOC minus Placebo + SOC
Statistical Analysis 2: Comparison: MK-6072 + SOC vs Placebo + SOC; Test type: Superiority or Other; p < 0.0001, Miettinen and Nurminen — [p-value comment as in outcome 1, analysis 1]; Adjusted Difference = 14.6, 95% CI 2-sided [7.7 to 21.4] — MK-6072 + SOC minus Placebo + SOC
Statistical Analysis 3: Comparison: MK-3415A + SOC vs MK-6072 + SOC; Test type: Superiority or Other; p = 0.9969, Miettinen and Nurminen — [p-value comment as in outcome 1, analysis 1]; Adjusted Difference = -9.4, 95% CI 2-sided [-16.1 to -2.7] — MK-3415A + SOC minus MK-6072 + SOC

3. Secondary Outcome: Percentage of Participants With CDI Recurrence in Those With Clinical Cure of the Initial CDI Episode
Description: CDI recurrence is defined as the development of a new episode of diarrhea (3 or more loose stools in 24 or fewer hours) and a positive lab stool test (local or central) for toxigenic C. difficile. Clinical cure is defined as no diarrhea [2 or fewer loose stools per 24 hours] for 2 consecutive days following completion of SOC therapy for the initial CDI episode in participants who received =< 14 day regimen.
Time Frame: 12 weeks
Population: Treated participants who achieved a clinical cure of the initial CDI episode.
Measure: Number; unit: Percentage of participants
Arm/Group | MK-3415A + SOC | MK-6072 + SOC | Placebo + SOC
Number analyzed (Participants) | 282 | 326 | 294
Percentage of participants | 20.6 | 19.0 | 33.0
Statistical Analysis 1: Comparison: MK-3415A + SOC vs Placebo + SOC; Test type: Superiority or Other; p = 0.0006, Miettinen and Nurminen — [p-value comment as in outcome 1, analysis 1]; Adjusted Difference = -11.9, 95% CI 2-sided [-19.0 to -4.7] — MK-3415A + SOC minus Placebo + SOC
Statistical Analysis 2: Comparison: MK-6072 + SOC vs Placebo + SOC; Test type: Superiority or Other; p < 0.0001, Miettinen and Nurminen — [p-value comment as in outcome 1, analysis 1]; Adjusted Difference = -13.7, 95% CI 2-sided [-20.4 to -6.9] — MK-6072 + SOC minus Placebo + SOC
Statistical Analysis 3: Comparison: MK-3415A + SOC vs MK-6072 + SOC; Test type: Superiority or Other; p = 0.6962, Miettinen and Nurminen — [p-value comment as in outcome 1, analysis 1]; Adjusted Difference = 1.6, 95% CI 2-sided [-4.6 to 8.0] — MK-3415A + SOC minus MK-6072 + SOC

4. Primary Outcome: Percentage of Participants With One or More Adverse Events During 4 Weeks Following Infusion Treatment
Description: An adverse event (AE) is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the medicinal product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the medicinal product, is also an adverse event.
Time Frame: Up to 4 weeks
Population: All Participants as Treated (APaT), based on the treatment actually received. One participant randomized to the MK- 3415A + SOC arm who was treated with MK-3415, but was not treated with MK-6072, was not analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | MK-3415A + SOC | MK-6072 + SOC | Placebo + SOC
Number analyzed (Participants) | 390 | 396 | 381
Percentage of participants | 57.4 | 58.1 | 60.4
Statistical Analysis 1: Comparison: MK-3415A + SOC vs Placebo + SOC; Test type: Superiority or Other; p = 0.408, Miettinen and Nurminen; Difference in Percentages = -2.9, 95% CI 2-sided [-9.8 to 4.0] — MK-3415A + SOC minus Placebo +SOC
Statistical Analysis 2: Comparison: MK-6072 + SOC vs Placebo + SOC; Test type: Superiority or Other; p = 0.517, Miettinen and Nurminen; Difference in Percentages = -2.3, 95% CI 2-sided [-9.2 to 4.6] — MK-6072 + SOC minus Placebo + SOC

5. Primary Outcome: Percentage of Participants With One or More Drug-related Adverse Events During 4 Weeks Following Infusion Treatment
Description: An adverse event (AE) is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the medicinal product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the medicinal product, is also an adverse event. A drug-related adverse event is determined by the investigator to be related to the drug.
Time Frame: Up to 4 weeks
Population: APaT based on the treatment actually received. One participant randomized to the MK-3415A + SOC arm who was treated with MK-3415, but was not treated with MK-6072, was not analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | MK-3415A + SOC | MK-6072 + SOC | Placebo + SOC
Number analyzed (Participants) | 390 | 396 | 381
Percentage of participants | 6.7 | 6.8 | 6.8
Statistical Analysis 1: Comparison: MK-3415A + SOC vs Placebo + SOC; Test type: Superiority or Other; p = 0.931, Miettinen and Nurminen; Difference in Percentages = -0.2, 95% CI 2-sided [-3.8 to 3.5] — MK-3415A + SOC minus Placebo + SOC
Statistical Analysis 2: Comparison: MK-6072 + SOC vs Placebo + SOC; Test type: Superiority or Other; p = 0.997, Miettinen and Nurminen; Difference in Percentages = 0.0, 95% CI 2-sided [-3.7 to 3.6] — MK-6072 + SOC minus Placebo + SOC

6. Primary Outcome: Percentage of Participants With One or More Serious Drug-related Adverse Events During 4 Weeks Following Infusion Treatment
Description: A serious adverse event (SAE) is any AE occurring at any dose or during any use of the medicinal product that results in death; or is life threatening; or results in a persistent or significant disability/incapacity; or results in or prolongs an existing inpatient hospitalization; or is a congenital anomaly/birth defect; or other important medical events. A serious drug-related adverse event is determined by the investigator to be related to the drug.
Time Frame: Up to 4 weeks
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | MK-3415A + SOC | MK-6072 + SOC | Placebo + SOC
Number analyzed (Participants) | 390 | 396 | 381
Percentage of participants | 0.8 | 0.0 | 0.3
Statistical Analysis 1: Comparison: MK-3415A + SOC vs Placebo + SOC; Test type: Superiority or Other; p = 0.328, Miettinen and Nurminen; Difference in Percentages = 0.5, 95% CI 2-sided [-0.8 to 2.0] — MK-3415A + SOC minus Placebo + SOC
Statistical Analysis 2: Comparison: MK-6072 + SOC vs Placebo + SOC; Test type: Superiority or Other; p = 0.308, Miettinen and Nurminen; Difference in Percentages = -0.3, 95% CI 2-sided [-1.5 to 0.7] — MK-6072 + SOC minus Placebo + SOC

7. Primary Outcome: Percentage of Participants Who Discontinued Study Medication Due to an Adverse Event During 4 Weeks Following Infusion Treatment
Description: as for outcome 4
Time Frame: Up to 4 weeks
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | MK-3415A + SOC | MK-6072 + SOC | Placebo + SOC
Number analyzed (Participants) | 390 | 396 | 381
Percentage of participants | 0 | 0 | 0
Statistical Analysis 1: Comparison: MK-3415A + SOC vs Placebo + SOC; Test type: Superiority or Other; p > 0.999, Miettinen and Nurminen; Difference in Percentages = 0.0, 95% CI 2-sided [-1.0 to 1.0] — MK-3415A + SOC minus Placebo + SOC
Statistical Analysis 2: Comparison: MK-6072 + SOC vs Placebo + SOC; Test type: Superiority or Other; p > 0.999, Miettinen and Nurminen; Difference in Percentages = 0.0, 95% CI 2-sided [-1.0 to 1.0] — MK-6072 + SOC minus Placebo + SOC

8. Primary Outcome: Percentage of Participants With One or More Infusion-specific Adverse Events on the Day of Infusion or the Day After Infusion
Description: as for outcome 4
Time Frame: Up to 24 hours
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | MK-3415A + SOC | MK-6072 + SOC | Placebo + SOC
Number analyzed (Participants) | 390 | 396 | 381
Percentage of participants | 7.2 | 8.8 | 7.6
Statistical Analysis 1: Comparison: MK-3415A + SOC vs Placebo + SOC; Test type: Superiority or Other; Difference in Percentages = -0.4, 95% CI 2-sided [-4.2 to 3.3] — MK-3415A + SOC minus Placebo + SOC
Statistical Analysis 2: Comparison: MK-6072 + SOC vs Placebo + SOC; Test type: Superiority or Other; Difference in Percentages = 1.2, 95% CI 2-sided [-2.7 to 5.2] — MK-6072 + SOC minus Placebo + SOC

9. Secondary Outcome: Percentage of Participants With CDI Recurrence in Those With a History of CDI in the 6 Months Prior to Enrollment
Description: as for outcome 3
Time Frame: 12 weeks
Population: Treated participants with a history of CDI in the past 6 months.
Measure: Number; unit: Percentage of participants
Arm/Group | MK-3415A + SOC | MK-6072 + SOC | Placebo + SOC
Number analyzed (Participants) | 104 | 113 | 110
Percentage of participants | 20.2 | 23.9 | 42.7

10. Secondary Outcome: Percentage of Participants With CDI Recurrence in Those With the 027 Ribotype
Description: CDI recurrence is defined as the development of a new episode of diarrhea (3 or more loose stools in 24 or fewer hours) and a positive lab stool test (local or central) for toxigenic C. difficile. Clinical cure is defined as no diarrhea [2 or fewer loose stools per 24 hours] for 2 consecutive days following completion of SOC therapy for the initial CDI episode in participants who received =< 14 day regimen. The 027 ribotype is a more virulent, epidemic strain responsible for several outbreaks of disease associated with an increased risk of severity and mortality.
Time Frame: 12 weeks
Population: Treated participants with the 027 ribotype
Measure: Number; unit: Percentage of participants
Arm/Group | MK-3415A + SOC | MK-6072 + SOC | Placebo + SOC
Number analyzed (Participants) | 39 | 43 | 64
Percentage of participants | 12.8 | 20.9 | 32.8

11. Secondary Outcome: Percentage of Participants With CDI Recurrence in Those With an Epidemic Strain
Description: CDI recurrence is defined as the development of a new episode of diarrhea (3 or more loose stools in 24 or fewer hours) and a positive lab stool test (local or central) for toxigenic C. difficile. Clinical cure is defined as no diarrhea [2 or fewer loose stools per 24 hours] for 2 consecutive days following completion of SOC therapy for the initial CDI episode in participants who received =< 14 day regimen. An epidemic strain includes ribotypes 027, 014, 002, 001, 106 or 020.
Time Frame: 12 weeks
Population: Treated participants with an epidemic strain
Measure: Number; unit: Percentage of participants
Arm/Group | MK-3415A + SOC | MK-6072 + SOC | Placebo + SOC
Number analyzed (Participants) | 116 | 102 | 127
Percentage of participants | 14.7 | 18.6 | 29.1

12. Secondary Outcome: Percentage of Participants With CDI Recurrence in Those With Clinically Severe CDI
Description: CDI recurrence is defined as the development of a new episode of diarrhea (3 or more loose stools in 24 or fewer hours) and a positive lab stool test (local or central) for toxigenic C. difficile. Clinical cure is defined as no diarrhea [2 or fewer loose stools per 24 hours] for 2 consecutive days following completion of SOC therapy for the initial CDI episode in participants who received =< 14 day regimen. Participants with clinically severe CDI have a Zar Score greater than or equal to 2 points based on the presence of 1 or more of the following: 1) age >60 years old (1 point); 2) body temperature >38.3°C (>100°F) (1 point); 3) albumin level ˂2.5 mg/dl (1 point); 4) peripheral white blood cell count >15,000 cells/mm^3 within 48 hours (1 point); 5) endoscopic evidence of pseudomembranous colitis (2 points); and 6) treatment in Intensive Care Unit (2 points).
Time Frame: 12 weeks
Population: Treated participants with clinically severe CDI
Measure: Number; unit: Percentage of participants
Arm/Group | MK-3415A + SOC | MK-6072 + SOC | Placebo + SOC
Number analyzed (Participants) | 80 | 55 | 65
Percentage of participants | 11.3 | 10.9 | 20.0

13. Secondary Outcome: Percentage of Participants With CDI Recurrence in Those 65 Years and Older
Description: as for outcome 3
Time Frame: 12 weeks
Population: Treated participants 65 years and older.
Measure: Number; unit: Percentage of participants
Arm/Group | MK-3415A + SOC | MK-6072 + SOC | Placebo + SOC
Number analyzed (Participants) | 241 | 205 | 206
Percentage of participants | 17.4 | 15.6 | 29.6

14. Secondary Outcome: Percentage of Participants With CDI Recurrence in Those With Compromised Immunity
Description: CDI recurrence is defined as the development of a new episode of diarrhea (3 or more loose stools in 24 or fewer hours) and a positive lab stool test (local or central) for toxigenic C. difficile. Clinical cure is defined as no diarrhea [2 or fewer loose stools per 24 hours] for 2 consecutive days following completion of SOC therapy for the initial CDI episode in participants who received =< 14 day regimen. Compromised immunity is an active hematological malignancy (including leukemia, lymphoma, multiple myeloma), an active malignancy requiring recent cytotoxic chemotherapy, receipt of a prior hematopoietic stem cell transplant, receipt of a prior solid organ transplant, asplenia, or neutropenia/pancytopenia due to other conditions.
Time Frame: 12 weeks
Population: Treated participants with compromised immunity
Measure: Number; unit: Percentage of participants
Arm/Group | MK-3415A + SOC | MK-6072 + SOC | Placebo + SOC
Number analyzed (Participants) | 85 | 91 | 61
Percentage of participants | 16.5 | 12.1 | 26.2

ADVERSE EVENTS:
Time Frame: Non-serious adverse events up to Day 28; serious adverse events up to Day 90
Description: Main Phase AEs were assessed Systematically: All Participants as Treated (APaT), based on the treatment actually received. One participant randomized to the MK-3415A + SOC arm was treated with MK-3415, but was not treated with MK-6072, is placed in his own arm for MK-3415 (not a randomized arm for this study).
  9-Month Extension AEs were not planned for collection; and were therefore assessed Non-systematically.
Groups:
- MK-3415A + SOC: Single IV infusion of 10 mg/kg MK 3415A + SOC for CDI
- MK-3415 + SOC: Single IV infusion of 10 mg/kg MK-3415 + SOC for CDI
Arm/Group | MK-3415A + SOC | MK-6072 + SOC | Placebo + SOC | MK-3415 + SOC | MK-3415A + SOC 9-ME | MK-6072 + SOC 9-ME | Placebo + SOC 9-ME
All-Cause Mortality (participants affected / at risk) | 31/390 | 25/396 | 33/381 | 1/1 | 2/112 | 5/100 | 2/83
Serious Adverse Events (participants affected / at risk) | 118/390 | 111/396 | 129/381 | 1/1 | 6/112 | 7/100 | 3/83
Other Adverse Events (participants affected / at risk) | 37/390 | 44/396 | 37/381 | 1/1 | 0/112 | 0/100 | 0/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | MK-3415A + SOC (N=390) | MK-6072 + SOC (N=396) | Placebo + SOC (N=381) | MK-3415 + SOC (N=1) | MK-3415A + SOC 9-ME (N=112) | MK-6072 + SOC 9-ME (N=100) | Placebo + SOC 9-ME (N=83)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac disorder (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 5 (5) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 5 (5) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prinzmetal angina (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blindness unilateral (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (5) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 7 (7) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 4 (4) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mesenteric artery thrombosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device breakage (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device malfunction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disuse syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug withdrawal syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic mass (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suprapubic pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bursitis infective staphylococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 13 (13) | 14 (15) | 28 (34) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cytomegalovirus viraemia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic foot infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungaemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HIV infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infective spondylitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningitis tuberculous (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 9 (9) | 5 (5) | 9 (9) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pseudomembranous colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 6 (7) | 13 (14) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 3 (3) | 1 (1) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 7 (7) | 9 (11) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriovenous fistula site haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Frostbite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural inflammation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood lactic acid increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shock hypoglycaemic (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medulloblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral T-cell lymphoma unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebellar haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Senile dementia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Status epilepticus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wernicke's encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephritic syndrome (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (4) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry gangrene (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shock (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Emphysematous cholecystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-3415A + SOC (N=390) | MK-6072 + SOC (N=396) | Placebo + SOC (N=381) | MK-3415 + SOC (N=1) | MK-3415A + SOC 9-ME (N=112) | MK-6072 + SOC 9-ME (N=100) | Placebo + SOC 9-ME (N=83)
Diarrhoea (Gastrointestinal disorders) | 17 (19) | 17 (18) | 21 (23) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 17 (17) | 23 (23) | 12 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 4 (5) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 1 (1) | 2 (3) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission.